CLINICAL TRIAL: NCT04589637
Title: Factors Influencing the Deterioration From Cognitive Decline of Normal Aging to Dementia Among Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: JUST20180229
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: A dearth of differential research exists regarding the determinants of mild cognitive impairment (MCI) and moderate cognitive impairment or dementia among nursing home residents. This study aimed to identify and examine the association between medical factors (number of comorbidities, hospitalization, disability, depression, frailty and quality of life) and moderate cognitive impairment or dementia in nursing homes residents.

Methods: A cross-sectional design was used in this study. Convenience sampling of 182 participants was conducted in nursing homes located in the central part of Jordan. Montreal cognitive assessment (MoCA) was used to screen both MCI and moderate cognitive impairment or dementia. Bivariate analysis, including t-test and ANOVA test, and logistic and linear regression models were used to examine and identify the medical factors associated with moderate cognitive impairment or dementia compared to mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Jordanian participants, aged 60 years and older, and living in nursing homes

Exclusion Criteria:

* neurological disorders, such as stroke or brain injury

Ages: 60 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Convenience sampling of 182 participants was used to obtain moderate size correlation (r = 0.35), given a power of 0.80, two-sided Type I error rate of p = 0.0167, based on nQuery calculation [16]. The participants were recruited from 5 holistic nursing homes, including private and public nursing homes, located in the center of Jordan. Inclusion criteria were as follows: Jordanian participants, aged 60 years and older, and living in nursing homes. Exclusion criteria were neurological disorders, such as stroke or brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
moderate cognitive impairment | May, 2018-May, 2019

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing homes, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kijowska V, Szczerbinska K. Prevalence of cognitive impairment among long-term care residents: a comparison between nursing homes and residential homes in Poland. Eur Geriatr Med. 2018 Aug;9(4):467-476. doi: 10.1007/s41999-018-0062-2. Epub 2018 May 16. PMID 34674486
- [Background] Hayajneh, A.A. , Ivanov, L.L. & Rababa, M. (2019). Jordanian Nursing Homes: Admission Policy Analysis. Global Journal of Health Science, 11 (6), 118-122.
- [Background] Janet D. Elashoff. nQuery Advisor Version 7.0 [software]. 2007: User's Guide. Los Angeles, CA
- [Background] The Montreal Cognitive Assessment (MoCA). What are the severity levels for the MoCA?. : Copyright 2019 Ziad Nasreddine MD. All rights reserved. Available from:: https://www.mocatest.org/faq/ [30August2020]
- [Background] Greenberg, S. Try this: the Geriatric Depression Scale (GDS). 2012: 4. The Hartford Institute for Geriatric Nursing, New York University, College of Nursing.
- [Background] Hayajneh, A. A. The Psychometric Properties of the Arabic Version of the Tilburg Frailty Indicator. Global Journal of Health Science. 2019: 11(9), 123-133. doi:10.5539/gjhs.v11n9p123
- [Background] Al-btoush, A. Relation between the Psychological Impact of Presbycusis and Hearing Handicap Inventory for the Elderly Using Screening Version in Jordan. Middle East Journal of Age and Ageing. 2012: 9(5), 23-25.
- [Background] Abdelmoneium, A.O. & Alharahsheh, S.T. Family Home Caregivers for Old Persons in the Arab Region: Perceived Challenges and Policy Implications. Open Journal of Social Sciences. 2016: 4, 151-164. http://dx.doi.org/10.4236/jss.2016.41019
- [Background] Arafa, Mohamed A., What's New in the Residential Care of the Elderly in the Arab and Islamic World? The Case of Egypt. Towards Human Rights in Residential Care for Older Persons: International Perspectives. 2015: (Chapter 2, Routledge, London & New York), Available at SSRN: https://ssrn.com/abstract=2710357
- [Background] Atif, M., Saleem, Q. & Scahill, S. Depression and mild cognitive impairment (MCI) among elderly patients with type 2 diabetes mellitus in Pakistan: possible determinants. Int J Diabetes Dev Ctries. 2018: 38, 312-320. https://doi.org/10.1007/s13410-017-0600-3
- [Background] Elliott, I. Poverty and Mental Health: A review to inform the Joseph Rowntree Foundation's Anti-Poverty Strategy. 2016: London: Mental Health Foundation.
- [Background] Mosti C.B., Rog L.A., Fink J.W. Differentiating Mild Cognitive Impairment and Cognitive Changes of Normal Aging. In: Ravdin L., Katzen H. (eds) Handbook on the Neuropsychology of Aging and Dementia. Clinical Handbooks in Neuropsychology. 2019. Springer, Cham
- [Result] Langa KM, Levine DA. The diagnosis and management of mild cognitive impairment: a clinical review. JAMA. 2014 Dec 17;312(23):2551-61. doi: 10.1001/jama.2014.13806. PMID 25514304
- [Result] Qarni T, Salardini A. A Multifactor Approach to Mild Cognitive Impairment. Semin Neurol. 2019 Apr;39(2):179-187. doi: 10.1055/s-0039-1678585. Epub 2019 Mar 29. PMID 30925611
- [Result] Ferreira AR, Dias CC, Fernandes L. Needs in Nursing Homes and Their Relation with Cognitive and Functional Decline, Behavioral and Psychological Symptoms. Front Aging Neurosci. 2016 Apr 21;8:72. doi: 10.3389/fnagi.2016.00072. eCollection 2016. PMID 27148044
- [Result] Bjork S, Juthberg C, Lindkvist M, Wimo A, Sandman PO, Winblad B, Edvardsson D. Exploring the prevalence and variance of cognitive impairment, pain, neuropsychiatric symptoms and ADL dependency among persons living in nursing homes; a cross-sectional study. BMC Geriatr. 2016 Aug 22;16(1):154. doi: 10.1186/s12877-016-0328-9. PMID 27549203
- [Result] Martin MD, Hancock GA, Richardson B, Simmons P, Katona C, Mullan E, Orrell M. An evaluation of needs in elderly continuing-care settings. Int Psychogeriatr. 2002 Dec;14(4):379-88. doi: 10.1017/s1041610202008578. PMID 12670059
- [Result] Ernsth Bravell M, Westerlind B, Midlov P, Ostgren CJ, Borgquist L, Lannering C, Molstad S. How to assess frailty and the need for care? Report from the Study of Health and Drugs in the Elderly (SHADES) in community dwellings in Sweden. Arch Gerontol Geriatr. 2011 Jul-Aug;53(1):40-5. doi: 10.1016/j.archger.2010.06.011. Epub 2010 Aug 3. PMID 20678818
- [Result] Gustafsson M, Sandman PO, Karlsson S, Isaksson U, Schneede J, Sjolander M, Lovheim H. Reduction in the use of potentially inappropriate drugs among old people living in geriatric care units between 2007 and 2013. Eur J Clin Pharmacol. 2015 Apr;71(4):507-15. doi: 10.1007/s00228-015-1825-z. Epub 2015 Feb 26. PMID 25716889
- [Result] Zheng L, Li G, Gao D, Wang S, Meng X, Wang C, Yuan H, Chen L. Cognitive frailty as a predictor of dementia among older adults: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2020 Mar-Apr;87:103997. doi: 10.1016/j.archger.2019.103997. Epub 2019 Dec 10. PMID 31846833
- [Result] Zuckerman H, Pan Z, Park C, Brietzke E, Musial N, Shariq AS, Iacobucci M, Yim SJ, Lui LMW, Rong C, McIntyre RS. Recognition and Treatment of Cognitive Dysfunction in Major Depressive Disorder. Front Psychiatry. 2018 Dec 4;9:655. doi: 10.3389/fpsyt.2018.00655. eCollection 2018. PMID 30564155
- [Result] Christiansen L, Sanmartin Berglund J, Lindberg C, Anderberg P, Skar L. Health-related quality of life and related factors among a sample of older people with cognitive impairment. Nurs Open. 2019 Mar 19;6(3):849-859. doi: 10.1002/nop2.265. eCollection 2019 Jul. PMID 31367408
- [Result] Park EY, Park SM, Kim JH. Psychometric properties of the geriatric quality of life-dementia in older adults with dementia or mild cognitive impairment living in nursing homes. BMC Geriatr. 2019 Oct 22;19(1):281. doi: 10.1186/s12877-019-1307-8. PMID 31640593
- [Result] Villeneuve R, Meillon C, Bergua V, Tabue-Teguo M, Amieva H. Influence of pre-admission factors on quality of life and adaptation in nursing home residents with dementia: the QOL-EHPAD study protocol. BMC Geriatr. 2020 Mar 6;20(1):92. doi: 10.1186/s12877-020-1434-2. PMID 32138680
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Sabbah I, Drouby N, Sabbah S, Retel-Rude N, Mercier M. Quality of life in rural and urban populations in Lebanon using SF-36 health survey. Health Qual Life Outcomes. 2003 Aug 6;1:30. doi: 10.1186/1477-7525-1-30. PMID 12952543
- [Result] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Result] Bani-Issa W, Almomani F, Eldeirawi K. Urinary incontinence among adult women with diabetes in Jordan: epidemiology, correlates and perceived impact on emotional and social well-being. J Clin Nurs. 2014 Sep;23(17-18):2451-60. doi: 10.1111/jocn.12392. Epub 2013 Sep 21. PMID 24112089
- [Result] Hussein S, Ismail M. Ageing and Elderly Care in the Arab Region: Policy Challenges and Opportunities. Ageing Int. 2017;42(3):274-289. doi: 10.1007/s12126-016-9244-8. Epub 2016 Apr 6. PMID 28890585
- [Result] Li W, Sun L, Li G, Xiao S. Prevalence, Influence Factors and Cognitive Characteristics of Mild Cognitive Impairment in Type 2 Diabetes Mellitus. Front Aging Neurosci. 2019 Jul 30;11:180. doi: 10.3389/fnagi.2019.00180. eCollection 2019. PMID 31417393
- [Result] Makizako H, Shimada H, Doi T, Tsutsumimoto K, Hotta R, Nakakubo S, Makino K, Suzuki T. Comorbid Mild Cognitive Impairment and Depressive Symptoms Predict Future Dementia in Community Older Adults: A 24-Month Follow-Up Longitudinal Study. J Alzheimers Dis. 2016 Oct 18;54(4):1473-1482. doi: 10.3233/JAD-160244. PMID 27589518
- [Result] Ma L. Depression, Anxiety, and Apathy in Mild Cognitive Impairment: Current Perspectives. Front Aging Neurosci. 2020 Jan 30;12:9. doi: 10.3389/fnagi.2020.00009. eCollection 2020. PMID 32082139
- [Result] Devanand DP, Pelton GH, D'Antonio K, Ciarleglio A, Scodes J, Andrews H, Lunsford J, Beyer JL, Petrella JR, Sneed J, Ciovacco M, Doraiswamy PM. Donepezil Treatment in Patients With Depression and Cognitive Impairment on Stable Antidepressant Treatment: A Randomized Controlled Trial. Am J Geriatr Psychiatry. 2018 Oct;26(10):1050-1060. doi: 10.1016/j.jagp.2018.05.008. Epub 2018 Jun 28. PMID 30037778
- [Result] Liu HY, Tsai WC, Chiu MJ, Tang LY, Lee HJ, Shyu YL. Mild cognitive impairment in combination with comorbid diabetes mellitus and hypertension is negatively associated with health-related quality of life among older persons in Taiwan. Qual Life Res. 2019 May;28(5):1281-1291. doi: 10.1007/s11136-019-02101-3. Epub 2019 Jan 11. PMID 30635850
- [Result] Chen TB, Yiao SY, Sun Y, Lee HJ, Yang SC, Chiu MJ, Chen TF, Lin KN, Tang LY, Lin CC, Wang PN. Comorbidity and dementia: A nationwide survey in Taiwan. PLoS One. 2017 Apr 12;12(4):e0175475. doi: 10.1371/journal.pone.0175475. eCollection 2017. PMID 28403222
- [Result] Solomon A, Dobranici L, Kareholt I, Tudose C, Lazarescu M. Comorbidity and the rate of cognitive decline in patients with Alzheimer dementia. Int J Geriatr Psychiatry. 2011 Dec;26(12):1244-51. doi: 10.1002/gps.2670. Epub 2011 Apr 16. PMID 21500282
- [Result] Stephan BC, Brayne C, Savva GM, Matthews FE; Medical Research Council Cognitive Function and Ageing Study. Occurrence of medical co-morbidity in mild cognitive impairment: implications for generalisation of MCI research. Age Ageing. 2011 Jul;40(4):501-7. doi: 10.1093/ageing/afr057. PMID 21673136
- [Result] Jacob L, Haro JM, Koyanagi A. Relationship between living alone and common mental disorders in the 1993, 2000 and 2007 National Psychiatric Morbidity Surveys. PLoS One. 2019 May 1;14(5):e0215182. doi: 10.1371/journal.pone.0215182. eCollection 2019. PMID 31042720
- [Result] Mathews SB, Arnold SE, Epperson CN. Hospitalization and cognitive decline: Can the nature of the relationship be deciphered? Am J Geriatr Psychiatry. 2014 May;22(5):465-80. doi: 10.1016/j.jagp.2012.08.012. Epub 2013 Feb 6. PMID 23567430
- [Result] Qin T, Yan M, Fu Z, Song Y, Lu W, Fu A, Yin P. Association between anemia and cognitive decline among Chinese middle-aged and elderly: evidence from the China health and retirement longitudinal study. BMC Geriatr. 2019 Nov 12;19(1):305. doi: 10.1186/s12877-019-1308-7. PMID 31718564
- [Result] Li M, Huang Y, Liu Z, Shen R, Chen H, Ma C, Zhang T, Li S, Prince M. The association between frailty and incidence of dementia in Beijing: findings from 10/66 dementia research group population-based cohort study. BMC Geriatr. 2020 Apr 15;20(1):138. doi: 10.1186/s12877-020-01539-2. PMID 32293307
- [Result] DeCarli C. Mild cognitive impairment: prevalence, prognosis, aetiology, and treatment. Lancet Neurol. 2003 Jan;2(1):15-21. doi: 10.1016/s1474-4422(03)00262-x. PMID 12849297
- [Result] Karrer M, Hirt J, Zeller A, Saxer S. What hinders and facilitates the implementation of nurse-led interventions in dementia care? A scoping review. BMC Geriatr. 2020 Apr 7;20(1):127. doi: 10.1186/s12877-020-01520-z. PMID 32264881
- [Result] Goossens B, Sevenants A, Declercq A, Van Audenhove C. 'We DECide optimized' - training nursing home staff in shared decision-making skills for advance care planning conversations in dementia care: protocol of a pretest-posttest cluster randomized trial. BMC Geriatr. 2019 Feb 4;19(1):33. doi: 10.1186/s12877-019-1044-z. PMID 30717700
- [Result] Zahirovic I, Torisson G, Wattmo C, Londos E. Psychotropic and anti-dementia treatment in elderly persons with clinical signs of dementia with Lewy bodies: a cross-sectional study in 40 nursing homes in Sweden. BMC Geriatr. 2018 Feb 17;18(1):50. doi: 10.1186/s12877-018-0740-4. PMID 29454305
- [Derived] Hayajneh AA, Rababa M, Alghwiri AA, Masha'al D. Factors influencing the deterioration from cognitive decline of normal aging to dementia among nursing home residents. BMC Geriatr. 2020 Nov 18;20(1):479. doi: 10.1186/s12877-020-01875-3. PMID 33208090